CLINICAL TRIAL: NCT02055248
Title: Study on Moebius Syndrome and Other Congenital Facial Weakness Disorders
Brief Title: Study on Moebius Syndrome and Congenital Facial Weakness Disorders
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Eye Institute (NEI) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Icahn School of Medicine at Mount Sinai (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140055; 14-HG-0055
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-14

CONDITIONS: Brain Disorders; Birth Defects; Craniofacial Differences
Keywords: Congenital Facial Weakness; Moebius; Cranial Nerve; Whole Exome Sequencing; Natural History
MeSH Terms: conditions — Brain Diseases; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Moebius or related syndromes and their family me: Subjects with Moebius or related syndromes and their family members and healthy volunteers.

SUMMARY:
Background:

- Moebius syndrome limits the ability to make facial expressions like smile, frown or blink - and move the eyes laterally. It can also cause speech, swallowing or breathing difficulties and affect parts of the body, such as the limbs, jaw, muscles, or the heart. Some individuals with Moebius can have intellectual impairment or behavior problems. Researchers want to study the clinical features of individuals with Moebius or related disorders and explore the genetic and/or environmental causes of these conditions.

Objective:

- To learn more about the genetics and clinical characteristics of Moebius syndrome and other Congenital Facial Weakness disorders.

Eligibility:

- People ages 2 to 80 years with congenital facial weakness, isolated or combined with other congenital anomalies, and their family members.

Design:

* Participants with Moebius syndrome or other congenital facial weakness disorder will be evaluated at the NIH Clinical Research Center over 3 to 5 days and undergo the following procedures:
* Medical and family history and physical examination, including body measurements and vital signs.
* Blood or saliva will be collected for genetic tests and to evaluate liver, kidney, heart and hormonal

functions.

* Eye examination, including having a video taken of their eyes moving.
* Hearing evaluation.
* Speech and language assessment, including swallowing studies.
* Dental exam.
* Detailed neurological evaluation, including electromyogram/nerve conduction and blink reflex study.
* Rehabilitation medicine evaluation, including muscle and tongue strength testing and assessment of balance.
* Neurocognitive and behavioral testing and questionnaires to assess quality of life and copying mechanisms.
* Imaging studies of their head, by magnetic resonance and diffusion tensor imaging -MRI/DTI. Participants

will lie on a table that slides into a metal cylinder that takes images of internal body structures using

magnets. Child participants may be sedated.

* Some adults may have additional X-rays of their head or limbs, if there are abnormal findings.
* Medical photographs of the face and affected body parts may be taken.
* Other specialized tests or consultations, as indicated.
* Participants can choose to have a skin biopsy taken.
* A follow-up visit will be offered to participants for review of genetic test findings and possibly additional clinical tests, as indicated.

Family members of the patients will have a medical and family history and physical examination. Blood or saliva will be obtained for genetic studies.

DETAILED DESCRIPTION:
This is a natural history study with a cross-sectional design of Moebius syndrome (MIM 157900), a heterogeneous developmental disorder defined as a congenital, non-progressive facial weakness with limited abduction of one or both eyes, often associated with additional features such as other cranial nerve dysfunction, craniofacial, skeletal and limb deformities, as well as intellectual or behavioral impairments. In this study we will attempt to characterize the clinical phenotype of Moebius and associated congenital facial weakness syndromes, collect thorough information on possible prenatal environmental exposures and use genetic studies, including whole exome sequencing, on DNA from patients and family members of patients to identify disease-causing genes. We will also conduct brain magnetic resonance- and diffusion tensor imaging- studies in these patients in order to explore brainstem and cranial nerve structure and associated white matter tract anomalies. Through this combined clinical, molecular and imaging approach, we anticipate that phenotype-genotype correlations will be revealed. These results will lead to new insights into the clinical definition of these conditions, molecular pathways, and potential networks involved in the pathogenesis of facial weakness and associated multisystem dysmorphogenesis. Our population will consist of patients, ages 2 to 80 years, inclusive of any gender, race, or ethnic group, with congenital facial palsy, isolated or combined with other congenital anomalies, and their families. We will continue to recruit approximately 24 probands each year, ages 2 to 80 years, inclusive of any gender, race, or ethnic group, and their parents and unaffected family members for a total of 72 patients/families. In most cases, patients will be referred through the Moebius Syndrome Foundation, a patient organization with a current membership of 2000 people in its database, 1400 of whom have been diagnosed with Moebius syndrome. Outcome measures will include the results from a battery of clinical evaluations, including ophthalmology, audiology, neurology, psychiatry, and rehabilitative medicine. Patients will also undergo neurocognitive and autism screening assessments, electromyography/nerve conduction, and blink reflex studies. Imaging and genetic studies will provide the most robust data for analysis in this study. A skin biopsy may be performed on some patients in order to culture fibroblasts for additional biochemical, cell biological, and molecular analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subject is 2-80 years, any gender, race or ethnic group, inclusive.
  2. Subject has a diagnosis of congenital facial palsy, isolated or combined with other congenital anomalies, based on MPIs review of prior medical records and interview with patient and/or patient physicians.
  3. Subject is a family member of a patient with a diagnosis of congenital facial palsy, isolated or combined with other congenital anomalies.
  4. Subject has the ability to travel to the NIH Clinical Center for admissions.
  5. Subject or subject s legal guardian is able to provide written informed consent.

EXCLUSION CRITERIA:

1. Subject has severe respiratory difficulties (i.e., requiring a tracheostomy or other assistive device to maintain respiration) or other disease manifestation that would interfere with the ability to comply with the requirements of this protocol and/or pose a severe anesthesia risk.
2. Subject has a psychiatric illness or neurological disease that would interfere with the ability to comply with the requirements of this protocol. This includes, but is not limited to, uncontrolled/untreated psychotic depression, bipolar disorder, schizophrenia, substance abuse or dependence, antisocial personality disorder, or panic disorder.
3. Subject shows evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, or gastrointestinal disease, or has a condition that requires immediate surgical intervention.
4. Subject is pregnant during the study.
5. Subject or subject s legal guardian is unable or unwilling to provide consent or assent.
6. The principal investigator may decline to enroll a patient for other reasons.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Moebius or related syndromes and their family members and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Employ genetic studies to study the molecular bases underlying congenital facial weakness syndromes. | One visit only
  Employ genetic studies, including comparative genomic hybridization, candidate gene testing and/or whole exome and genome sequencing to study the molecular bases underlying these syndromes. Our hypothesis is that disease-causing mutations will be present in the proteincoding regions of the genome, as germline or somatic mutations. In the future whole genome sequencing may be considered.
Characterize the phenotype of patients with typical Moebius syndrome | One visit only
  To characterize the phenotype of patients with typical Moebius syndrome, defined as uni- or bilateral facial and uni- or bilateral abducens nerve palsy and patients with atypical Moebius-like phenotypes that include facial weakness, including Moebius-Poland, Moebius-Robin or Moebius-Kallmann syndromes, Carey-Fineman-Ziter syndrome, Hereditary Congenital Facial Paresis (HCFP), oculoauriculovertebral dysplasia (Goldenhar syndrome), among others, and determine the prevalence of associated malformations. Our primary hypothesis is that oculomotor, neuromuscular, skeletal or imaging endophenotypes will help categorize the various groups more accurately and inform subsequent genetic studies.

SECONDARY OUTCOMES:
Obtain brain-imaging studies including DTI/tractography | one time only
  Obtain brain-imaging studies including DTI/tractography in a large cohort of patients with congenital malformations associated with facial weakness to explore anomalies in brain and brainstem structure and associated white matter anomalies and fiber tract connectivity, together with a careful delineation of patients' neurocognitive andbehavioral phenotype. Results from this distinct developmental disorder will be compared to data from normal children and children with non-syndromic autism.
Study the neurocognitive, behavioral, and quality of life outcomes of individuals with congenital facial weakness | one time only
  Study the neurocognitive, behavioral, and quality of life outcomes of individuals with these syndromes, and provide proper genetic counseling about management, prognosis, and recurrence risk to affected families

CONTACTS AND LOCATIONS:
Overall Officials: Eirini Manoli, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Di Gioia SA, Connors S, Matsunami N, Cannavino J, Rose MF, Gilette NM, Artoni P, de Macena Sobreira NL, Chan WM, Webb BD, Robson CD, Cheng L, Van Ryzin C, Ramirez-Martinez A, Mohassel P, Leppert M, Scholand MB, Grunseich C, Ferreira CR, Hartman T, Hayes IM, Morgan T, Markie DM, Fagiolini M, Swift A, Chines PS, Speck-Martins CE, Collins FS, Jabs EW, Bonnemann CG, Olson EN; Moebius Syndrome Research Consortium; Carey JC, Robertson SP, Manoli I, Engle EC. A defect in myoblast fusion underlies Carey-Fineman-Ziter syndrome. Nat Commun. 2017 Jul 6;8:16077. doi: 10.1038/ncomms16077. PMID 28681861
- [Background] Telegrafi A, Webb BD, Robbins SM, Speck-Martins CE, FitzPatrick D, Fleming L, Redett R, Dufke A, Houge G, van Harssel JJT, Verloes A, Robles A, Manoli I, Engle EC; Moebius Syndrome Research Consortium; Jabs EW, Valle D, Carey J, Hoover-Fong JE, Sobreira NLM. Identification of STAC3 variants in non-Native American families with overlapping features of Carey-Fineman-Ziter syndrome and Moebius syndrome. Am J Med Genet A. 2017 Oct;173(10):2763-2771. doi: 10.1002/ajmg.a.38375. Epub 2017 Aug 4. PMID 28777491
- [Background] Webb BD, Shaaban S, Gaspar H, Cunha LF, Schubert CR, Hao K, Robson CD, Chan WM, Andrews C, MacKinnon S, Oystreck DT, Hunter DG, Iacovelli AJ, Ye X, Camminady A, Engle EC, Jabs EW. HOXB1 founder mutation in humans recapitulates the phenotype of Hoxb1-/- mice. Am J Hum Genet. 2012 Jul 13;91(1):171-9. doi: 10.1016/j.ajhg.2012.05.018. Epub 2012 Jul 5. PMID 22770981
- [Derived] Japee S, Jordan J, Licht J, Lokey S; Moebius Syndrome Research Consortium; Chen G, Snow J, Jabs EW, Webb BD, Engle EC, Manoli I, Baker C, Ungerleider LG. Inability to move one's face dampens facial expression perception. Cortex. 2023 Dec;169:35-49. doi: 10.1016/j.cortex.2023.08.014. Epub 2023 Sep 30. PMID 37852041
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-HG-0055.html